CLINICAL TRIAL: NCT03017235
Title: A Randomized, Assessor-Blinded, Multi-Center Study Investigating the Efficacy, Safety, and Tolerability of Sodium Picosulfate, Magnesium Oxide and Anhydrous Citric Acid Oral Solution Versus Sodium Picosulfate, Magnesium Oxide and Anhydrous Citric Acid Powder for Oral Solution (PREPOPIK®) for Colon Cleansing in Preparation for Colonoscopy
Brief Title: A Study Comparing the Sodium Picosulfate, Magnesium Oxide and Anhydrous Citric Acid Oral Solution With PREPOPIK® for Colon Cleansing in Preparation for Colonoscopy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ferring Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 000253
Record Dates: First submitted 2017-01-09; First posted 2017-01-11 (Estimated); Results first posted 2018-11-14 (Actual); Last update posted 2018-11-14 (Actual); Status verified 2018-10

CONDITIONS: Bowel Preparation
MeSH Terms: interventions — picosulfate sodium; Magnesium Oxide; Citric Acid

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- NaP/MC Oral Solution (Experimental): Sodium Picosulfate, Magnesium Oxide and Anhydrous Citric Acid (NaP/MC) Oral Solution
  Interventions: Drug: Sodium Picosulfate, Magnesium Oxide and Anhydrous Citric Acid Oral Solution
- PREPOPIK® (Active Comparator)
  Interventions: Drug: Sodium Picosulfate, Magnesium Oxide and Anhydrous Citric Powder

INTERVENTIONS:
Drug: Sodium Picosulfate, Magnesium Oxide and Anhydrous Citric Acid Oral Solution — Supplied as two 160 mL ready-to-drink bottles, per subject, without further reconstitution, before administration.
  Arms: NaP/MC Oral Solution
Drug: Sodium Picosulfate, Magnesium Oxide and Anhydrous Citric Powder — Supplied as two sachets per subject. Subjects will be instructed to reconstitute the medication by combining the contents of one packet with approximately five (5) ounces of cold water and stirring for two to three minutes.
  Other Names: PREPOPIK®; PicoPrep®
  Arms: PREPOPIK®

SUMMARY:
The purpose of this study is to compare the Sodium Picosulfate, Magnesium Oxide and Anhydrous Citric Acid Oral Solution with PREPOPIK® for colon cleansing in adult subjects undergoing colonoscopy.

ELIGIBILITY:
Inclusion Criteria:

* Male or non-pregnant female subjects aged 18 to 80 years, inclusive, being scheduled to undergo elective colonoscopy
* Females of childbearing potential must agree to use an adequate contraception during the course of the trial. Accepted forms of contraception are: i.e., implants, injectables, hormonal intrauterine device, combined hormonal contraceptives, sexual abstinence, and vasectomized sexual partner. Premenopausal women who are of childbearing potential must have a negative serum pregnancy test result at screening and a negative urine pregnancy test result at randomization prior to colonoscopy. In the case of oral contraceptive use, women should have been taking the same pill consistently for a minimum of twelve (12) weeks before taking study medication. Sterilized or postmenopausal women may also participate. Women are considered to be postmenopausal and are not considered to be of childbearing potential if they have had twelve (12) months of natural (spontaneous) amenorrhea with an appropriate clinical profile (e.g. age appropriate, history of vasomotor symptoms) or have had surgical bilateral oophorectomy (with or without hysterectomy) or tubal ligation.
* An average of at least 3 spontaneous bowel movements per week for one month prior to the colonoscopy

Exclusion Criteria:

* Known or suspected gastrointestinal obstruction, perforation, ileus, or gastric retention
* Acute intestinal or gastric ulceration
* Severe acute inflammatory bowel disease (IBD), toxic colitis, or toxic megacolon
* Undergoing colonoscopy for foreign body removal or decompression
* Reduced level of consciousness or inability to swallow without aspiration
* Any prior colorectal surgery, excluding appendectomy, hemorrhoid surgery, or prior endoscopic procedures
* Upper gastrointestinal surgery (gastrectomy, gastric banding, gastric by-pass)
* Uncontrolled angina and/or myocardial infarction (MI) within last three months, congestive heart failure (CHF), uncontrolled hypertension, or ascites
* Severely reduced renal function (<30 mL/min/1.73 m2)
* Pregnant or lactating women
* Any clinically relevant abnormal findings in medical history, physical examination, vital signs, ECG, clinical chemistry, hematology, coagulation, or urinalysis at Screening Visit 1
* Rhabdomyolysis
* Chronic nausea and vomiting
* Hypermagnesemia
* Undergoing treatment with Lithium

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 917 (Actual)
Dates: Start 2017-02-20 (Actual); Primary Completion 2017-09-15 (Actual); Study Completion 2017-10-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Development Support, Study Director — Ferring Pharmaceuticals
Locations (14):
- United States (12):
  - Clinical Research Associates, Huntsville, Alabama
  - Associated Gastroenterology Medical Group, Anaheim, California
  - GW Research, Inc., Chula Vista, California
  - Precision Research Institute, San Diego, California
  - Connecticut Clinical Research Foundation, Bristol, Connecticut
  - Florida Clinical Research Group, Clearwater, Florida
  - Nature Coast Clinical Research, Inverness, Florida
  - Long Island Gastrointestinal Research Group LLC, Great Neck, New York
  - Kinston Medical Specialists, PA, Kinston, North Carolina
  - Wake Research Associates, LLC, Raleigh, North Carolina
  - Hillmont GI, Flourtown, Pennsylvania
  - Advanced Research Institute, Ogden, Utah
- Canada (2):
  - Hotel Dieu Hospital, Kingston
  - Canadian Phase Onward, Inc., Toronto

REFERENCES:
- [Derived] Mankaney GN, Ando M, Dahdal DN, Burke CA. Safety and efficacy of sodium picosulfate, magnesium oxide, and citric acid bowel preparation in patients with baseline renal impairment or diabetes: subanalysis of a randomized, controlled trial. Therap Adv Gastroenterol. 2021 Jun 28;14:17562848211024458. doi: 10.1177/17562848211024458. eCollection 2021. PMID 34262611
- [Derived] Hookey L, Bertiger G, Johnson KL 2nd, Boules M, Ando M, Dahdal DN. Efficacy, safety, and tolerability of a ready-to-drink bowel preparation in overweight and obese adults: subanalysis by body mass index from a phase III, assessor-blinded study. Therap Adv Gastroenterol. 2020 Apr 9;13:1756284820910050. doi: 10.1177/1756284820910050. eCollection 2020. PMID 32313553
- [Derived] Hookey L, Bertiger G, Johnson KL, Boules M, Ando M, Dahdal DN. Efficacy, safety, and tolerability of a ready-to-drink bowel preparation: subanalysis by age from a phase III, assessor-blinded study. Therap Adv Gastroenterol. 2020 Feb 7;13:1756284820902878. doi: 10.1177/1756284820902878. eCollection 2020. PMID 32095161
- [Derived] Hookey L, Bertiger G, Lee Johnson K 2nd, Ayala J, Seifu Y, Brogadir SP. Efficacy and safety of a ready-to-drink bowel preparation for colonoscopy: a randomized, controlled, non-inferiority trial. Therap Adv Gastroenterol. 2019 May 19;12:1756284819851510. doi: 10.1177/1756284819851510. eCollection 2019. PMID 31205487

RESULTS

PARTICIPANT FLOW:
Groups:
- NaP/MC Oral Solution: Sodium Picosulfate, Magnesium Oxide and Anhydrous Citric Acid (NaP/MC) Oral Solution
  Supplied as two 160 mL ready-to-drink bottles, per subject without further reconstitution, before administration.
  Split dose regimen: Subjects began treatment (first dose) the evening before colonoscopy between 5:00 PM and 9:00 PM, and completed treatment (second dose) the following day, at least 5 hours, but no more than 9 hours, prior to the colonoscopy.
- PREPOPIK®: Sodium Picosulfate, Magnesium Oxide and Anhydrous Citric Powder: Supplied as two packets per subject.
  Split dose regimen :Subjects will be instructed to reconstitute the medication by combining the contents of one packet with approximately five (5) ounces of cold water and stirring for two to three minutes.
  Subjects began treatment (first dose) the evening before colonoscopy between 5:00 PM and 9:00 PM, and completed treatment (second dose) the following day, at least 5 hours, but no more than 9 hours, prior to the colonoscopy.
Period: Overall Study
Arm/Group | NaP/MC Oral Solution | PREPOPIK®
Started | 456 | 461
Completed | 444 | 447
Not Completed | 12 | 14
Not completed — Withdrawal by Subject | 4 | 3
Not completed — Lost to Follow-up | 2 | 7
Not completed — Adverse Event | 0 | 1
Not completed — Protocol Violation | 2 | 1
Not completed — Cancer, emergency, allergy, active UTI | 4 | 2

BASELINE CHARACTERISTICS:
Population: Modified intention-to-treat (mITT) was considered as the main analysis set. mITT was defined as all ITT subjects who received at least 1 dose of treatment. The mITT analysis set was analyzed according to randomized treatment.
Groups:
- NaP/MC Oral Solution: Sodium Picosulfate, Magnesium Oxide and Anhydrous Citric Acid (NaP/MC) Oral Solution
  Sodium Picosulfate, Magnesium Oxide and Anhydrous Citric Acid Oral Solution: Supplied as ready-to-drink without further reconstitution before administration
- PREPOPIK®: Sodium Picosulfate, Magnesium Oxide and Anhydrous Citric Powder: Supplied as two packets per subject. Subjects will be instructed to reconstitute the medication by combining the contents of one packet with approximately five (5) ounces of cold water and stirring for two to three minutes.
- Total: Total of all reporting groups
Arm/Group | NaP/MC Oral Solution | PREPOPIK® | Total
Number analyzed (Participants) | 448 | 453 | 901
Age, Continuous [Mean (Standard Deviation); unit: Years] | 57.2 (11.04) | 57.1 (10.85) | 57.2 (10.94)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 252 | 250 | 502
  Male | 196 | 203 | 399
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 68 | 71 | 139
  Not Hispanic or Latino | 380 | 381 | 761
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 13 | 5 | 18
  Native Hawaiian or Other Pacific Islander | 1 | 1 | 2
  Black or African American | 49 | 41 | 90
  White | 376 | 394 | 770
  More than one race | 2 | 2 | 4
  Unknown or Not Reported | 7 | 9 | 16
Child-bearing potential [Number; unit: Participants]
  Child bearing potential | 252 | 250 | 502
  Yes | 49 | 47 | 96
  No | 203 | 203 | 406

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects Classified as a Responder Defined by "Excellent" or "Good"
Description: The efficacy of overall colon cleansing in terms of responders was measured by a blinded endoscopist using the Modified Aronchick Scale. Modified Aronchick scale is a 4-point scale that grades colon cleansing as Excellent (>90% of mucosa seen, mostly liquid stool, minimal suctioning needed for adequate visualization), Good (>90% of mucosa seen, mostly liquid stool, significant suctioning needed for adequate visualization), Fair (>90% of mucosa seen, mixture of liquid and semisolid stool, could be suctioned and/or washed) or Inadequate (<90% of mucosa seen, mixture of semisolid and solid stool which could not be suctioned or washed).The participant is considered to be a responder if overall colon cleansing is "excellent" or "good" on this 4-point scale.
Time Frame: During colonoscopy procedure (5-9 hours after completed treatment)
Population: The primary efficacy analysis was conducted for the mITT analysis set and was defined as all ITT subjects who received at least 1 dose of treatment. The mITT analysis set was analyzed according to randomized treatment.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- NaP/MC Oral Solution: Sodium Picosulfate, Magnesium Oxide and Anhydrous Citric Acid (NaP/MC) Oral Solution
  Supplied as two 160 mL ready-to-drink bottles, per subject without further reconstitution, before administration.
Arm/Group | NaP/MC Oral Solution | PREPOPIK®
Number analyzed (Participants) | 448 | 453
Percentage of participants | 87.7 [84.3 to 90.6] | 81.5 [77.6 to 84.9]
Statistical Analysis 1: Comparison: NaP/MC Oral Solution vs PREPOPIK®; Difference in the percentage of subjects on NaP/MC or PREPOPIK (NaP/MC - PREPOPIK); Test type: Non-Inferiority — The NI margin for the difference between treatments (NaP/MC Oral Solution minus PREPOPIK) was pre-specified at -8% (absolute). If NI was demonstrated for both the primary efficacy endpoint and the secondary efficacy endpoint for the right colon, and if the lower bound of the CI was above 0%, then superiority was declared for the primary endpoint. Thus, the pre-specified superiority analysis was conducted at a one-sided significance level of 2.5%; p = 0.0067, Weighted Percentage Difference — The above p-value was calculated for superiority and was based on the stratified percentage difference test, where the stratification weight is based on Cochran-Mantel-Haenszel-weight; CIs (treatment difference) were calculated using stratified (by site) percentage difference where, weights= Cochran-Mantel-Haenszel weights for site; Difference in percentage = 6.3, 95% CI 2-sided [1.8 to 10.9]; Lower limit of 95% CI > 0% for the primary efficacy endpoint combined with outcome of secondary efficacy endpoint for the right colon allowed for superiority analysis

2. Secondary Outcome: Percentage of Subjects Classified as a Responder Defined by a Score ≥2 in the Right Segment of the Colon
Description: The percentage of subjects classified as responders, defined by a Boston Bowel Preparation Scale (BBPS) score ≥2 in the right segment of the colon was determined.
  The BBPS scale:
  0= Unprepared colon segment with mucosa not seen due to solid stool that cannot be cleared; 1= Portion of mucosa of the colon segment seen, but other areas of the colon segment not well seen due to staining, residual stool, and/or opaque liquid; 2= Minor amount of residual staining, small fragments of stool and/or opaque liquid, but mucosa of colon segment seen well; 3= Entire mucosa of colon segment seen well with no residual staining, small fragments of stool or opaque liquid.
Time Frame: During colonoscopy procedure (5-9 hours after completed treatment)
Population: The efficacy analysis was conducted for the mITT analysis set and was defined as all ITT subjects who received at least 1 dose of treatment. The mITT analysis set was analyzed according to randomized treatment.
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | NaP/MC Oral Solution | PREPOPIK®
Number analyzed (Participants) | 448 | 453
Percentage of subjects | 94.2 [91.6 to 96.2] | 89.6 [86.4 to 92.3]
Statistical Analysis 1: Comparison: NaP/MC Oral Solution vs PREPOPIK®; Difference in the percentage of subjects on NaP/MC or PREPOPIK (NaP/MC - PREPOPIK); Test type: Non-Inferiority — If the lower limit of the 95% CI was greater than the margin (-8%), the null hypothesis was rejected and NaP/MC Oral Solution was claimed as non-inferior to PREPOPIK with respect to right colon cleansing in preparation for colonoscopy; p = 0.0099, Weighted Percentage Difference — The p-value was calculated for superiority and was based on the stratified percentage difference test, where the stratification weight is based on Cochran-Mantel-Haenszel-weight; [statistical method as in outcome 1, analysis 1]; Difference in percentage = 4.6, 95% CI 2-sided [1.1 to 8.0]

3. Secondary Outcome: Percentage of Subjects Classified as a Responder Defined by a Score ≥2 in the Transverse Segment of the Colon
Description: The percentage of subjects classified as responders, defined by a Boston Bowel Preparation Scale (BBPS) score ≥2 in the transverse segment of the colon was determined.
  The BBPS scale:
  0= Unprepared colon segment with mucosa not seen due to solid stool that cannot be cleared; 1= Portion of mucosa of the colon segment seen, but other areas of the colon segment not well seen due to staining, residual stool, and/or opaque liquid; 2= Minor amount of residual staining, small fragments of stool and/or opaque liquid, but mucosa of colon segment seen well; 3= Entire mucosa of colon segment seen well with no residual staining, small fragments of stool or opaque liquid.
Time Frame: During colonoscopy procedure (5-9 hours after completed treatment)
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | NaP/MC Oral Solution | PREPOPIK®
Number analyzed (Participants) | 448 | 453
Percentage of subjects | 96.0 [93.7 to 97.6] | 94.0 [91.4 to 96.0]
Statistical Analysis 1: Comparison: NaP/MC Oral Solution vs PREPOPIK®; Difference in percentage of subjects on NaP/MC Oral Solution or PREPOPIK® (NaP/MC - PREPOPIK); Test type: Non-Inferiority — [test comment as in outcome 2, analysis 1]; p = 0.1781, Weighted Percentage Difference — The above p-value was tested for superiority and was based on the stratified percentage difference test, where the stratification weight is based on Cochran Mantel Haenszel weight; [statistical method as in outcome 1, analysis 1]; Difference in percentage = 1.9, 95% CI 2-sided [-0.9 to 4.7]

4. Secondary Outcome: Percentage of Subjects Classified as a Responder Defined by a Score ≥2 in the Left Segment of the Colon
Description: The percentage of subjects classified as responders, defined by a Boston Bowel Preparation Scale (BBPS) score ≥2 in the left segment of the colon was determined.
  The BBPS scale:
  0= Unprepared colon segment with mucosa not seen due to solid stool that cannot be cleared; 1= Portion of mucosa of the colon segment seen, but other areas of the colon segment not well seen due to staining, residual stool, and/or opaque liquid; 2= Minor amount of residual staining, small fragments of stool and/or opaque liquid, but mucosa of colon segment seen well; 3= Entire mucosa of colon segment seen well with no residual staining, small fragments of stool or opaque liquid.
Time Frame: During colonoscopy procedure (5-9 hours after completed treatment)
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | NaP/MC Oral Solution | PREPOPIK®
Number analyzed (Participants) | 448 | 453
Percentage of subjects | 94.6 [92.1 to 96.5] | 91.2 [88.2 to 93.6]
Statistical Analysis 1: Comparison: NaP/MC Oral Solution vs PREPOPIK®; Difference in percentage of subjects on NaP/MC Oral Solution or PREPOPIK® (NaP/MC-PREPOPIK®); Test type: Non-Inferiority — If the lower limit of the 95% CI was greater than the margin (-8%), the null hypothesis was rejected and NaP/MC Oral Solution was claimed as non-inferior to PREPOPIK with respect to colon cleansing in preparation for colonoscopy; p = 0.0391, Weighted Percentage Difference — The above p-value was for superiority and was based on the stratified percentage difference, where the stratification weight is based on Cochran-Mantel-Haenszel weight; [statistical method as in outcome 1, analysis 1]; Difference in percentage = 3.5, 95% CI 2-sided [0.2 to 6.7]

5. Secondary Outcome: Frequency of Each Category on the Subject Tolerability Questionnaire (How Many Bowel Movements Did You Have in the Week Prior to Starting Colon Preparation?)
Description: Subject tolerability and satisfaction with the bowel cleansing preparation were assessed by the validated Mayo Clinic Bowel Prep Tolerability Questionnaire. This simple, comprehensive questionnaire, developed to evaluate the tolerability of various types of bowel preparations, was administered to the subject at Visit 3 prior to the colonoscopy procedure.
Time Frame: During colonoscopy procedure (5-9 hours after completed treatment)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | NaP/MC Oral Solution | PREPOPIK®
Number analyzed (Participants) | 448 | 453
Participants
  ≤3/week | 63 | 47
  4 to 8/week | 264 | 299
  ≥9/week | 120 | 105
  Response not provided | 0 | 1
  Not applicable | 1 | 1

6. Secondary Outcome: Frequency of Each Category on the Subject Tolerability Questionnaire (How Much Bowel Preparation Was Left in Bottle After Drinking it?)
Description: as for outcome 5
Time Frame: During colonoscopy procedure (5-9 hours after completed treatment)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | NaP/MC Oral Solution | PREPOPIK®
Number analyzed (Participants) | 448 | 453
Participants
  <25% | 443 | 448
  25% - 50% | 1 | 1
  50% - 75% | 0 | 2
  ≥75% | 1 | 0
  Response not provided | 2 | 1
  Not applicable | 1 | 1

7. Secondary Outcome: Frequency of Each Category on the Subject Tolerability Questionnaire (Was the Bowel Preparation Tolerable?)
Description: as for outcome 5
Time Frame: During colonoscopy procedure (5-9 hours after completed treatment)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | NaP/MC Oral Solution | PREPOPIK®
Number analyzed (Participants) | 448 | 453
Participants
  Easy to acceptable | 400 | 433
  Somewhat difficult | 41 | 17
  Very difficult | 4 | 1
  Unacceptable | 2 | 1
  Not applicable | 1 | 1

8. Secondary Outcome: Frequency of Each Category on the Subject Tolerability Questionnaire (How Willing Are You to Use This Preparation in the Future?)
Description: as for outcome 5
Time Frame: During colonoscopy procedure (5-9 hours after completed treatment)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | NaP/MC Oral Solution | PREPOPIK®
Number analyzed (Participants) | 448 | 453
Participants
  Not willing at all | 11 | 6
  Somewhat willing | 75 | 38
  Mostly willing | 361 | 408
  Not applicable | 1 | 1

9. Secondary Outcome: Frequency of Each Category on the Subject Tolerability Questionnaire (If Difficulties Existed, Were They Due to Your Current Health Status?)
Description: Subject tolerability and satisfaction with the bowel cleansing preparation were assessed by the validated Mayo Clinic Bowel Prep Tolerability Questionnaire. This simple, comprehensive questionnaire, developed to evaluate the tolerability of various types of bowel preparations, was administered to the subject at Visit 3 prior to the colonoscopy procedure. Subjects in response to questions could provide multiple response if applicable.
Time Frame: During colonoscopy procedure (5-9 hours after completed treatment)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | NaP/MC Oral Solution | PREPOPIK®
Number analyzed (Participants) | 448 | 453
Participants
  Yes | 11 | 8
  No | 104 | 93
  No difficulties | 310 | 320
  No health issues | 84 | 109
  Response not provided | 0 | 3

10. Secondary Outcome: Frequency of Each Category on the Subject Tolerability Questionnaire (How Bothered Were You During Bowel Prep by Bad Taste in Mouth?)
Description: as for outcome 5
Time Frame: During colonoscopy procedure (5-9 hours after completed treatment)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | NaP/MC Oral Solution | PREPOPIK®
Number analyzed (Participants) | 448 | 453
Participants
  Not bothered-Mildly bothered | 371 | 426
  Moderately bothered | 63 | 22
  Severely bothered | 11 | 2
  No response | 1 | 3
  Not applicable | 2 | 0

11. Secondary Outcome: Frequency of Each Category on the Subject Tolerability Questionnaire (How Bothered Were You During Bowel Prep by Gastric Fullness?)
Description: as for outcome 5
Time Frame: During colonoscopy procedure (5-9 hours after completed treatment)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | NaP/MC Oral Solution | PREPOPIK®
Number analyzed (Participants) | 448 | 453
Participants
  Not bothered-Mildly bothered | 382 | 387
  Moderately bothered | 53 | 57
  Severely bothered | 10 | 6
  No response | 2 | 3
  Not applicable | 1 | 0

12. Secondary Outcome: Frequency of Each Category on the Subject Tolerability Questionnaire (How Bothered Were You During Bowel Prep by Lack of Sleep From Excessive Bathroom Trips?)
Description: as for outcome 5
Time Frame: During colonoscopy procedure (5-9 hours after completed treatment)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | NaP/MC Oral Solution | PREPOPIK®
Number analyzed (Participants) | 448 | 453
Participants
  Not bothered-Mildly bothered | 335 | 328
  Moderately bothered | 86 | 85
  Severely bothered | 25 | 37
  No response | 1 | 3
  Not applicable | 1 | 0

13. Secondary Outcome: Frequency of Each Category on the Subject Tolerability Questionnaire (How Bothered Were You During Bowel Prep by Nausea, Vomiting?)
Description: as for outcome 5
Time Frame: During colonoscopy procedure (5-9 hours after completed treatment)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | NaP/MC Oral Solution | PREPOPIK®
Number analyzed (Participants) | 448 | 453
Participants
  Not bothered-Mildly bothered | 416 | 435
  Moderately bothered | 23 | 11
  Severely bothered | 6 | 2
  No response | 2 | 4
  Not applicable | 1 | 0

14. Secondary Outcome: Frequency of Each Category on the Subject Tolerability Questionnaire (How Bothered Were You During Bowel Prep by Bloating/Abdominal Distension/Gas?)
Description: as for outcome 5
Time Frame: During colonoscopy procedure (5-9 hours after completed treatment)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | NaP/MC Oral Solution | PREPOPIK®
Number analyzed (Participants) | 448 | 453
Participants
  Not bothered-Mildly bothered | 403 | 402
  Moderately bothered | 35 | 40
  Severely bothered | 7 | 6
  No response | 2 | 4
  Not applicable | 1 | 1

15. Secondary Outcome: Frequency of Each Category on the Subject Tolerability Questionnaire (How Bothered Were You During Bowel Prep by Abdominal Pain/Cramps?)
Description: as for outcome 5
Time Frame: During colonoscopy procedure (5-9 hours after completed treatment)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | NaP/MC Oral Solution | PREPOPIK®
Number analyzed (Participants) | 448 | 453
Participants
  Not bothered-Mildly bothered | 427 | 432
  Moderately bothered | 15 | 15
  Severely bothered | 3 | 3
  No response | 1 | 2
  Not applicable | 2 | 1

16. Secondary Outcome: Frequency of Each Category on the Subject Tolerability Questionnaire (How Bothered Were You During Bowel Prep by Headache?)
Description: as for outcome 5
Time Frame: During colonoscopy procedure (5-9 hours after completed treatment)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | NaP/MC Oral Solution | PREPOPIK®
Number analyzed (Participants) | 448 | 453
Participants
  Not bothered-Mildly bothered | 396 | 396
  Moderately bothered | 38 | 47
  Severely bothered | 13 | 7
  No response | 0 | 2
  Not applicable | 1 | 1

17. Secondary Outcome: Frequency of Each Category on the Subject Tolerability Questionnaire (Was This Your First Colonoscopy?)
Description: as for outcome 5
Time Frame: During colonoscopy procedure (5-9 hours after completed treatment)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | NaP/MC Oral Solution | PREPOPIK®
Number analyzed (Participants) | 448 | 453
Participants
  No | 261 | 281
  Yes | 185 | 171
  Response not provided | 1 | 2
  Not applicable | 1 | 0

18. Secondary Outcome: Frequency of Each Category on the Subject Tolerability Questionnaire (Previous Bowel Preparation)
Description: as for outcome 5
Time Frame: During colonoscopy procedure (5-9 hours after completed treatment)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | NaP/MC Oral Solution | PREPOPIK®
Number analyzed (Participants) | 448 | 453
Participants
  GoLytely | 56 | 52
  Moviprep | 14 | 17
  MiraLax | 20 | 20
  Other | 34 | 39
  Do not remember | 137 | 53

19. Secondary Outcome: Frequency of Each Category on the Subject Tolerability Questionnaire (Tolerability Compared to Previous Bowel Prepreparations)
Description: as for outcome 5
Time Frame: During colonoscopy procedure (5-9 hours after completed treatment)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | NaP/MC Oral Solution | PREPOPIK®
Number analyzed (Participants) | 448 | 453
Participants
  Worse than before | 5 | 5
  About the same as before | 62 | 67
  Better than before | 190 | 209
  Response not provided | 4 | 0

20. Secondary Outcome: Percentage of Treatment-emergent Adverse Events(AEs)
Description: Collected as any AE that begins during the treatment period defined as the period during which a subject receives IMP. All endoscopy findings were reported as AEs while cancers/malignancies detected on endoscopy were reported as SAEs.
Time Frame: From baseline (screening) up to day 28 after colonoscopy
Population: The Safety analysis set comprised all subjects who received any amount of study medication. The Safety analysis set was analyzed according to the actual treatment received
Measure: Number; unit: Percentage of adverse events
Arm/Group | NaP/MC Oral Solution | PREPOPIK®
Number analyzed (Participants) | 448 | 453
Percentage of adverse events | 84.4 | 84.8

21. Secondary Outcome: Clinically Significant Changes in Vital Signs
Description: Blood pressure and pulse will be measured after at least 5 minutes of rest in supine position and after 3 minutes in standing position
Time Frame: From baseline (screening) up to day 28 after colonoscopy
Population: as for outcome 20
Measure: Count of Participants; unit: Participants
Arm/Group | NaP/MC Oral Solution | PREPOPIK®
Number analyzed (Participants) | 448 | 453
Participants
  Hypertension | 0 | 4
  Orthostatic hypotension | 1 | 2
  Blood pressure increased | 2 | 0
  Hypotension | 1 | 1

22. Secondary Outcome: Clinically Significant Changes in Electrocardiogram (ECG)
Description: Measured by standard 12-lead ECG. At each visit when an ECG was done, the investigator reviewed and initialed the tracing, which was then stored with the subject's source documents. The baseline ECG performed at the Screening Visit was reviewed for major abnormalities before dosing.
Time Frame: At baseline (screening), on the day of colonoscopy, 1-2 days after colonoscopy, 7 days after colonoscopy and 28 days after colonoscopy
Population: as for outcome 20
Measure: Count of Participants; unit: Participants
Arm/Group | NaP/MC Oral Solution | PREPOPIK®
Number analyzed (Participants) | 448 | 453
Participants
  Bradycardia | 3 | 0
  Bundle branch block left | 0 | 2
  Extrasystoles | 0 | 2
  Ventricular extrasystoles | 2 | 0
  Atrial fibrillation | 1 | 0
  Bundle branch block right | 1 | 0
  Palpitations | 1 | 0
  Sinus bradycardia | 0 | 1
  Tachycardia | 0 | 1
  Cardiac murmur | 1 | 0

23. Secondary Outcome: Clinically Significant Changes in Laboratory Values
Description: Rated by the investigator based on out of range laboratory values
Time Frame: as for outcome 22
Population: as for outcome 20
Measure: Count of Participants; unit: Participants
Arm/Group | NaP/MC Oral Solution | PREPOPIK®
Number analyzed (Participants) | 448 | 453
Participants
  Hematology: Anaemia | 1 | 1
  Hematology: Leukopenia | 1 | 0
  Hematology: Lymphocytosis | 0 | 1
  Hematology: Neutropenia | 1 | 0
  Hematology: Normocytic anaemia | 1 | 0
  Hemotology: Platelet count decreased | 0 | 1
  Clinical Chemistry: Hypermagnesaemia | 9 | 23
  Clinical chemistry:Blood bicarbonate decreased | 6 | 3
  Clinical chemistry: Hypokalemia | 4 | 0
  Clinical chemistry: Hyperglycaemia | 2 | 1
  Clinical chemistry: Hypoglycaemia | 3 | 0
  Clinical chemistry: Hyperkalaemia | 0 | 2
  Clinical chemistry: Hypomagnasaemia | 2 | 0
  Clinical chemistry: Blood creatinine increased | 0 | 1
  Clinical chemistry: Blood potassium decreased | 1 | 0
  Clinical chemistry: Hypochloraemia | 0 | 1
  Clinical chemistry: Hyperbilirubinaemia | 0 | 1
  Urinalysis | 0 | 0

ADVERSE EVENTS:
Time Frame: From baseline (screening) upto 28 days after colonoscopy.
Groups:
- NaP/MC Oral Solution: Sodium Picosulfate, Magnesium Oxide and Anhydrous Citric Acid (NaP/MC) Oral Solution
  Supplied as two 160 mL ready-to-drink bottles per subject without further reconstitution before administration.
- PREPOPIK®: Sodium Picosulfate, Magnesium Oxide and Anhydrous Citric Powder
  Supplied as two packets per subject. Subjects will be instructed to reconstitute the medication by combining the contents of one packet with approximately five (5) ounces of cold water and stirring for two to three minutes.
Arm/Group | NaP/MC Oral Solution | PREPOPIK®
All-Cause Mortality (participants affected / at risk) | 0/448 | 0/453
Serious Adverse Events (participants affected / at risk) | 9/448 | 6/453
Other Adverse Events (participants affected / at risk) | 378/448 | 384/453
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NaP/MC Oral Solution (N=448) | PREPOPIK® (N=453)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Ascites (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 0 (0) | 1 (1)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4) | 0 (0)
Rectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Breast cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Carcinoid tumour of the gastrointestinal tract (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NaP/MC Oral Solution (N=448) | PREPOPIK® (N=453)
Haemorrhoids (Gastrointestinal disorders) | 150 (162) | 155 (167)
Large intestine polyp (Gastrointestinal disorders) | 93 (157) | 105 (181)
Diverticulum intestinal (Gastrointestinal disorders) | 70 (75) | 70 (73)
Diverticulum (Gastrointestinal disorders) | 64 (64) | 59 (59)
Investigations (Infections and infestations) | 25 (26) | 23 (26)
Hypermagnesaemia (Metabolism and nutrition disorders) | 9 (9) | 23 (26)
Colon adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 133 (237) | 128 (211)
Infections and infestations (Infections and infestations) | 27 (29) | 35 (35)
Nervous system disorders (Nervous system disorders) | 27 (27) | 30 (34)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI is that the sponsor can review the draft manuscript prior to publication and can request delay of publication where any contents are deemed patentable by the sponsor or confidential to the sponsor. Comments will be given within four weeks from receipt of the draft manuscript. Additional time may be required to allow Ferring to seek patent protection of the invention.

DOCUMENTS (2):
  • Study Protocol (2017-01-25): https://cdn.clinicaltrials.gov/large-docs/35/NCT03017235/Prot_000.pdf
  • Statistical Analysis Plan (2017-12-01): https://cdn.clinicaltrials.gov/large-docs/35/NCT03017235/SAP_001.pdf